CLINICAL TRIAL: NCT04962919
Title: Survival Outcomes in Metastatic Prostate Cancer in the Brazilian Population - Analysis of Individual Characteristics and Treatment Modalities in Different National Health Institutions.
Acronym: LACOG 1818
Status: Active, not recruiting | Type: Observational
Sponsor: Latin American Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: LACOG 1818
Record Dates: First submitted 2021-06-24; First posted 2021-07-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Prostatic Neoplasms, Castration-Resistant
Keywords: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Public institution: Castration-resistant metastatic prostate cancer diagnosed between January 2014 and December 2017
- Private institution: Castration-resistant metastatic prostate cancer diagnosed between January 2014 and December 2017

SUMMARY:
Survival outcomes in metastatic prostate cancer in the population Brazilian - analysis of individual characteristics and modalities of treatment in different national health institutions

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of castration-resistant metastatic prostate cancer diagnosed in the period between January 2014 and December 2017.

Exclusion Criteria:

* Diagnosis of localized or locally advanced or metastatic disease sensitive to castration;
* Patients with medical records filled with incomplete data that make it impossible to evaluate the treatment received.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of castration-resistant metastatic prostate cancer diagnosed in the period between January 2014 and December 2017.
Sampling Method: Non-Probability Sample
Enrollment: 584 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2025-05-07 (Estimated); Study Completion 2025-05-07 (Estimated)

PRIMARY OUTCOMES:
Describe cause-specific survival in patients with castration-resistant prostate cancer in different institutions in Brazil. | December of 2017

SECONDARY OUTCOMES:
To describe the sociodemographic characteristics of patients with castration-resistant metastatic prostate cancer in Brazil; | December of 2017
To describe comorbidities of patients with castration-resistant metastatic prostate cancer in Brazil; | December of 2017
To describe the clinicopathological characteristics of patients with metastatic castration-resistant prostate cancer in Brazil; | December of 2017
To compare overall survival among patients with castration-resistant metastatic prostate cancer treated in the SUS and in the private network; | December of 2017
To compare the treatments performed by patients with castration-resistant metastatic prostate cancer in the SUS and in the private network; | December of 2017
To describe the rates of skeletal-related complications | December of 2017
To describe the rate of admissions | December of 2017
To describe the number of lines of treatment that patients have undergone | December of 2017
To describe the presence or absence of treatments bone-directed | December of 2017

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Cotait Maluf, Principal Investigator — Latin American Cooperative Oncology Group
Locations (8):
- Brazil (8):
  - CPO Pucrs, Porto Alegre, Rio Grande do Sul
  - Centro de Estudos e Pesquisas de Hematologia e Oncologia - CEPHO, Santo André, São Paulo
  - Sírio Libanês, São Paulo, São Paulo
  - Centro Paulista de Oncologia, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo
  - BP - A Beneficência Portuguesa de São Paulo, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São Paulo - Hospital Central, São Paulo
  - A.C.Camargo Cancer Center, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided